CLINICAL TRIAL: NCT03163706
Title: Evaluation of Stroop Effect in Patients With Schizophrenia
Acronym: STROOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHU-330; 2014-A00957-40 (Other: 2014-A00957-40)
Record Dates: First submitted 2017-05-11; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Stroop effect; Semantic conflict; Response conflict
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Masking Description: Open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schizophrenia patients (Experimental): Patients with DSM-5 criteria of schizophrenia
  Interventions: Behavioral: Modified Stroop effect
- Control group (Other): Control, no schizophrenia
  Interventions: Behavioral: Modified Stroop effect

INTERVENTIONS:
Behavioral: Modified Stroop effect — to assess whether attention deficits and executive functions in patients with schizophrenia are general (semantic and response conflict) or specific (semantic or response conflict).

SUMMARY:
The main objective of this study is to assess whether attention deficits and executive functions in patients with schizophrenia are general (semantic and response conflict) or specific (semantic or response conflict).

DETAILED DESCRIPTION:
First, participants will receive six categories of stimuli presented in a classical way: (1) incongruous stimulus classical (BLUE written in green for example); (2) associated incongruous stimuli (SKY written in green for example); (3) conventional congruent stimuli (BLUE written in blue for example); (4) associated congruent stimuli (SKY written in blue for example); (5) neutral words (BRIDGE written in green for example); And (6) neutral stimulus (XXXX written in green for example).

In a second step (after a 5 minute break), they will receive these six categories of stimuli, but only half will be presented in a classic way and the other half will be presented in order to attract attention as in Augustinova and Ferrand 2007). To do this, in (1) incongruous stimuli classical like BLUE, a single letter (like B for example) will be colored in green for example and the rest of the word (LUE) will appear in gray); In (2) incongruous stimuli associated as SKY, only K for example will be green and the rest of the word will appear in gray); In (3) conventional congruent stimuli such as BLUE, only B for example will be written in blue and the rest of the word will appear in gray); In (4) associated congruent stimuli such as SKY only K for example will be written in blue and the rest of the word will appear in gray); In (5) neutral words like BRIDGE, only D will be colored in green for example and the rest of the word will appear in gray; And finally, in (6) neutral stimuli like XXXX, only one X will be colored in green for example and the rest of the X will appear in gray.

The task will be to name the color of each word (by stating the color verbally) as quickly and correctly as possible, while ignoring the written word. In this experiment, we will measure the time taken to denominate the color (in milliseconds) as well as the percentages of incorrect answers.

The first step allows to determine the stroop effect and the second the semantic conflict.

ELIGIBILITY:
Inclusion Criteria:

For both:

* MMSE score greater than or equal to, 22 if no grade ; 23 if study certificate or CAP or college without patent ; 25 if patent or school without the tray ; 26 or more when bin
* IQ ≥ 75 (fNART)
* Lextale score ≥ 28
* Age: between 18 and 45 years

For patients :

* DSM-5 criteria of schizophrenia
* Patients followed as outpatients,
* Age of onset of the disease less than 40 years,
* Patients whose disease has stabilized: no changes psychotropic treatment for at least 1 month
* Not more of a benzodiazepine,
* Patients on protection of justice or not,

For controls :

* Matched for sex to patient
* Age-matched (+/- 3 years) to patient
* Matched for IQ (score fNART +/- 10% to patients
* Matched for Lextale score+/- 10% to patients

Exclusion Criteria:

For patients :

* Any other comorbid psychiatric diagnosis of Axis I DSM-5
* Extrapyramidal syndrome or tardive dyskinesia (AIMS score <2 BARS score <2 and score Simpson and Angus <3)
* Calgary depression scale ≥ 6
* Current or past addiction to all toxic substances (including alcohol and cannabis) except tobacco.
* Current or past use of all toxic consumption (excluding alcohol, tobacco and cannabis).
* Use of alcohol or cannabis before the age of 15 years
* Alcohol abuse in the past 6 months.
* Cannabis abuse in the past 6 months and cannabis use in the last 3 months.
* Patients with impaired vision or hearing preventing the realization of the tests.

For controls:

* Any psychiatric diagnosis according to DSM-5, including addictions (excluding tobacco)
* Score HADS Anxiety ≥ 8 and Depression ≥ 8
* SCL90R: global severity score GSI> 0.33 for women and> 0.27 for men, or score diversity PST symptoms> 18.49 for men and> 21.97 for women or score of degree of discomfort PSDI> 1.27 for men and> 1.3 for women, scoring in the subscale Psychotic Features> 0.
* Presence of a personality disorder at PDQ4 +
* Head injuries, brain injuries or diseases,
* vision or hearing problems preventing the realization of the tests.
* Current or past addiction to all toxic substances (including alcohol and cannabis) except tobacco.
* Current or past use of all toxic consumption (excluding alcohol, tobacco and cannabis).
* Long-term Anticholinergic treatment.
* Related to the first degree diagnosed with a psychotic disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-09-21 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Semantic conflict in stroop test | at day 1
  The stroop effect consists of the semantic and the response conflict. In patients with schizophrenia, the stroop effect is longer than in controls. By comparing the stroop effect and the semantic conflict between patients and controls, we can determine whether the slowing observed in patients is due to a general slowdown (semantic and response conflict) or specific slowness (semantic or response conflict).

SECONDARY OUTCOMES:
Response conflict in stroop test | at day 1
  The stroop effect consists of the semantic and the response conflict. In patients with schizophrenia, the stroop effect is longer than in controls. Response conflict (time in milliseconds) is obtained by subtracting the semantic conflict (time in milliseconds obtained in the second step of the protocol) from the stroop effect (time in milliseconds obtained in the first step of the protocol).
  Therefore, we can determine whether the slowing observed in patients is due to a general slowdown (semantic and response conflict) or specific slowness (semantic or response conflict).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France